CLINICAL TRIAL: NCT04514887
Title: Intraoperative Mild Hyperventilation as an Intervention to Decrease the Incidence of Postoperative Shoulder Pain After Gastric Sleeve Bypass Surgery
Brief Title: Mild Intraoperative Hyperventilation to Decrease Post-op. Shoulder Pain After LSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Adel Mefleh Abdallah Bataineh, Principal Investigator, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 56/124/2019
Record Dates: First submitted 2020-08-09; First posted 2020-08-17 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Laparoscopic Gastric Sleeve Surgery; ASA-I and II Risk Class Patients; Same Surgeon

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the anesthetist administering the anesthesia and mechanical ventilation is Awarem of the arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild Hyperventilation (Experimental): In this study arm, patients were mildly hyperventilated intraoperatively so their end-tidal CO2 levels are brought down to 30-32 mmHg.
  Interventions: Other: mild intraoperative hyperventilation
- Control (No Intervention): In this study arm patients' ventilation is managed according to guidelines with end-tidal CO2 levels kept in the normal range of 35-40 mm Hg

INTERVENTIONS:
Other: mild intraoperative hyperventilation — Intraoperative mechanical ventilation of patients was adjusted so that end-tidal CO2 readings lie between 30-32 mmHg
  Arms: Mild Hyperventilation

SUMMARY:
Shoulder pain is common after laparoscopic surgeries. multiple maneuvers are in use to decrease its incidence with variable results. This study aims to investigate the effect of mild hyperventilation to an End-tidal CO2 level of 30-32 mmHg on the occurrence of postoperative shoulder pain. This is carried out through a comparison of the incidence of postoperative shoulder pain an intervention group to that in a control one with a normal End Tidal CO2 35-40 mmHg). controlling for all other variables.

DETAILED DESCRIPTION:
This novel technique is based on the theory that shoulder pain is caused by diaphragmatic irritation by CO2 during laparoscopic surgery. The investigators postulate that lowering the CO2 level in the plasma, will lower tissue CO2 level in the diaphragm and decrease the hypothesized irritation. In this study, patients will be divided into an interventional group which will receive mild intraoperative hyperventilation determined by an End-Tidal CO2 level of 30-32 mm Hg and a control group in which End Tidal CO2 is kept at normal levels (35-40 mmHg). All other intraoperative factors will be standardized for all patients. Patients will be followed up postoperatively and asked whether the participants developed shoulder pain as a primary study outcome. The pain will be recorded in terms of severity, site, and position, and any associations (Nausea and vomiting). Appropriate statistical tests will be used to check for any significant effects of the technique.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* No mental illnesses
* American Society of Anesthesiologists (ASA) class I&II,
* Patients undergoing laparoscopic sleeve gastrectomy.
* No previous intrabdominal surgeries.

Exclusion Criteria:

* ASA class >II,
* previous abdominal surgeries.
* mental illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-06-16 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Postoperative shoulder Pain | 3 months
  patient complaining of left of right shoulder pain after laparoscopic sleeve gastrectomy will be evaluated using numerical rating scale, were zero indicates no pain at all, and 10 indicates most severe pain the patient has ever had.

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | 3 months
  The development of nausea and vomiting among patients after laparoscopic sleeve gastrectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Adel M Bataineh, MD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- King Abdullah Teaching Hospital, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sao CH, Chan-Tiopianco M, Chung KC, Chen YJ, Horng HC, Lee WL, Wang PH. Pain after laparoscopic surgery: Focus on shoulder-tip pain after gynecological laparoscopic surgery. J Chin Med Assoc. 2019 Nov;82(11):819-826. doi: 10.1097/JCMA.0000000000000190. PMID 31517775
- [Background] Donatsky AM, Bjerrum F, Gogenur I. Surgical techniques to minimize shoulder pain after laparoscopic cholecystectomy. A systematic review. Surg Endosc. 2013 Jul;27(7):2275-82. doi: 10.1007/s00464-012-2759-5. Epub 2013 Jan 24. PMID 23340814
- [Background] Pergialiotis V, Vlachos DE, Kontzoglou K, Perrea D, Vlachos GD. Pulmonary recruitment maneuver to reduce pain after laparoscopy: a meta-analysis of randomized controlled trials. Surg Endosc. 2015 Aug;29(8):2101-8. doi: 10.1007/s00464-014-3934-7. Epub 2014 Nov 1. PMID 25361653
- [Background] Phelps P, Cakmakkaya OS, Apfel CC, Radke OC. A simple clinical maneuver to reduce laparoscopy-induced shoulder pain: a randomized controlled trial. Obstet Gynecol. 2008 May;111(5):1155-60. doi: 10.1097/AOG.0b013e31816e34b4. PMID 18448749